CLINICAL TRIAL: NCT06906354
Title: The Effect of Intrabronchial Therapy With Gentamycin and Dexamethason After Bronchoscopic Airway Clearance in Exacerbation of Bronchiectasis
Brief Title: Airway Clearance by Fiberoptic Bronchoscopy in Bronchiectasis Followed by Gentamicin and Dexamethason Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: bronchiectasis FOB
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Bronchiectasis Adult; Bronchiectasis With Acute Exacerbation
Keywords: bronchoscopy; bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: Fiberoptic Airway Clearance in Bronchiectasis Exacerbation and Gentamicin-Dexamethason Injection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fiberoptic bronchoscopy in one group (Active Comparator): Airway Clearance by Fiberoptic Bronchoscopy in Bronchiectasis Followed by Gentamicin and Dexamethason Injection
  Interventions: Procedure: Airway Clearance by Fiberoptic Bronchoscopy in Bronchiectasis Followed by Gentamicin and Dexamethason Injection

INTERVENTIONS:
Procedure: Airway Clearance by Fiberoptic Bronchoscopy in Bronchiectasis Followed by Gentamicin and Dexamethason Injection — Airway Clearance by Fiberoptic Bronchoscopy in Bronchiectasis Followed by Gentamicin and Dexamethason Injection

SUMMARY:
Fiberoptic Bronchoscopic Removal of Secretions and Antibiotic Injection

DETAILED DESCRIPTION:
fiberoptic bronchoscopic injection of dexamethason and gentamicin after airway clearance

ELIGIBILITY:
Inclusion Criteria:

1- Adult subjects. 2- Male and female subjects are enrolled. 3- patients with NCFB confirmed by chest high-resolution computed tomography (HRCT) 4- patients needing antibiotic treatment at the hospital due to exacerbation 5- Patients who underwent AC by bronchoscopy at the hospital.

-

Exclusion Criteria:

1- Uncooperative subjects. 2- Unwilling to participate. 3- Inability to lie on the back with raised arms over the head for HRCT. 4- Presence of cystic pulmonary fibrosis; 5- Patients with active pulmonary tuberculosis; 6- Those awaiting surgery; 7- Patients who underwent interventional therapy for hemoptysis; those with allergic bronchopulmonary aspergillosis (ABPA); 8- Patients who did not undergo bronchoscopy for different reasons or combined with lung cancer.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Dyspnea Borg Scale | one month
  improvement in the scale of dyspnea before and after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: mohamed sabry Eltarhony, lecturer, Principal Investigator — Alexandria University
Locations (1):
- Chest Department -Faculty of Medicine, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i will do it after being accepted from the ethics committee

REFERENCES:
- See also: bronchoscopy in bronchiectasis — https://pubmed.ncbi.nlm.nih.gov/30545985/
- See also: fiberoptic bronchoscopy in bronchiectasis — https://pubmed.ncbi.nlm.nih.gov/17482984/
- Available data/document: Study Protocol: msabry776@yahoo.com — https://pubmed.ncbi.nlm.nih.gov/17482984/ — very good